CLINICAL TRIAL: NCT06564350
Title: Digitalization of Measuring Physical Performance
Status: Completed | Type: Observational
Sponsor: Yale University (Other)
Responsible Party: Sponsor
Other Study IDs: 2000034742
Record Dates: First submitted 2024-08-19; First posted 2024-08-21 (Actual); Last update posted 2024-08-21 (Actual); Status verified 2024-08

CONDITIONS: Physical Performance

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Modified Physical Performance test (MPPT): Participants will perform MPPT with and without the wearable seonsors.
  Interventions: Device: IMU (Inertial Measurement Unit) sensors

INTERVENTIONS:
Device: IMU (Inertial Measurement Unit) sensors — IMU sensors track an object's acceleration and angular velocity over time and do not emit any electromagnetic fields or radiation. They use tiny masses and springs to measure the acceleration, as well as Hall effect materials to measure the magnetic fields. The force sensor changes its electric resistor value based on the force applied to the sensor surface.

SUMMARY:
Investigators will test the validity and reproducibility of the measurement of motor performance using wearables and the correlation of this measurement with function and mobility.

DETAILED DESCRIPTION:
The primary objective of this study is to determine whether the digital measurement of physical performance delivers more accurate and more consistent results than the current traditional measurement of physical performance done by rehabilitation therapists in the rehabilitation patient population.

The primary outcome of this study is to check the correlation between the traditional rehabilitation test scores of Modified Physical Performance test (MPPT), and measured values via the wearables.

The MPPT consists of sub-tasks, which are part of standard physical and occupational therapy evaluation and treatment in the inpatient rehabilitation setting. During the therapy session 4-8 sensors will be applied to participant over their clothing. As the participant performs various subtasks of MPPT the wearable sensors will provide measurements. At the same time the physical or occupational therapist will do measurements on the same subtasks in the traditional way which is based on observation and time to complete a task. A gaming component is being added to the sub task of balance. For the subtask of balance the participant will be wearing the wearable sensor for balance and at the same time will be looking at an animation on a screen. The participant will try to control a moving object on the gaming screen with their balance. The scoring on the gaming component also gives a digital score of the participants balance. In this case of the balance subtask the physical therapist will do the measurement of the balance in the traditional way with observation and time to complete the subtask. The performance of all subtasks by the participants, will be with a licensed physical therapist as part of the routine physical therapy evaluation and treatment session.

The schedule of digital measurements of physical performance by wearable sensors for each participant will be on THREE occasions as follows:

1. During the initial physical and occupational therapy evaluation session -approximately 1 hour duration
2. During a physical/occupational therapy session within 1 -2 weeks after the initial evaluation - approximately 1 hour duration
3. During a physical/occupational therapy session within 1-2 weeks after the second evaluation or at time of discharge - approximately 1 hour duration

ELIGIBILITY:
Inclusion Criteria:

* Participants can stand with or without an assistive device with or without assistance form another person/s
* Participants can walk with or without an assistive device with or without assistance from another person/s
* Participants are able to memorize easy tasks, and able to follow instructions e.g., standing up or walking until a certain location in the room

Exclusion Criteria:

* Participants who are not cleared physically or medically to participate in standard acute inpatient rehabilitation therapies by the rehabilitation physician
* Not able to memorize easy tasks, e.g., standing up or walking until a certain location in the room
* One or more leg/feet amputated

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants are patients admitted to acute inpatient rehabilitation unit for rehabilitation who are able to stand and walk with or without an assistive device.
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2023-07-27 (Actual); Primary Completion 2023-08-04 (Actual); Study Completion 2023-08-11 (Actual)

PRIMARY OUTCOMES:
Digitalized scores of physical performance | up to 5 weeks
  A percentage score, which determines how well a participant can do motor tasks for strength, balance, mobility, range of motion and tasks of activities of daily life. Computer software will be used to evaluate the test score of the patient using information from the wearable sensors. The resulting score will be evaluated with the help of a Regression Machine Learning Algorithm. These results will be compared to the assessment and scoring of physical performance by rehabilitation therapists that is based on observation. Higher percentage indicates better performance.

CONTACTS AND LOCATIONS:
Overall Officials: Rummana Aslam, MD, Principal Investigator — Yale University
Locations (1):
- Yale New Haven Hospital Rehabilitation and Wellness center, New Haven, Connecticut, United States